CLINICAL TRIAL: NCT01140581
Title: A Randomized, International, Multi-center, Open-label Study to Document Optimal Timing of Initiation of Dronedarone Treatment After Conversion With Loading Dose of Amiodarone in Patients With Persistent Atrial Fibrillation Requiring Conversion of AF.
Brief Title: Optimal Timing of Dronedarone Initiation After Conversion in Patients With Persistent Atrial Fibrillation
Acronym: ARTEMIS Load
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRONE_C_03668; 2009-016818-24 (EudraCT Number)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Amiodarone 600 mg daily for 1 week then 400 mg daily for 1 week then 200 mg daily for 2 weeks followed by dronedarone 400 mg twice daily for 8 weeks
  Interventions: Drug: DRONEDARONE
- Group B (Experimental): Amiodarone 600 mg daily for 1 week then 400 mg daily for 1 week then 200 mg daily for 2 weeks. Two weeks wash-out followed by dronedarone 400 mg twice daily for 6 weeks
  Interventions: Drug: DRONEDARONE
- Group C (Experimental): Amiodarone 600 mg daily for 1 week then 400 mg daily for 1 week then 200 mg daily for 2 weeks. Four weeks wash-out followed by dronedarone 400 mg twice daily for 4 weeks
  Interventions: Drug: DRONEDARONE

INTERVENTIONS:
Drug: DRONEDARONE — Pharmaceutical form: tablet Route of administration: oral Dose regimen: 400 mg

SUMMARY:
Primary Objective:

- Evaluate the rate of Atrial Fibrillation (AF) recurrences one month after randomization according to different timings of initiation of dronedarone.

Secondary Objective:

* Evaluate the rate of AF recurrences two months after randomization.
* Assess the safety of the change from amiodarone to dronedarone
* Assess dronedarone safety
* Explore dronedarone and its active metabolite plasma level (in a subset of countries)
* Explore potential Pharmacokinetic (PK) interaction between dronedarone and amiodarone (in a subset of countries)

ELIGIBILITY:
Inclusion criteria:

Screening:

* Persistent AF for more than 72 hours (documented by an ECG taken within the last 72 hours) for whom cardioversion, anti-arrhythmic treatment and anticoagulation treatment are indicated in the opinion of the Investigator
* Naive of amiodarone treatment in the last three months
* QTc Bazett < 500 ms on 12-lead ECG,
* At least one cardiovascular risk factor (i.e. age > 70, hypertension, diabetes, prior cerebrovascular disease or left atrial diameter >= 50 mm

Randomization:

* Outpatient and Inpatients (except patients hospitalized during screening period for SAE)
* Sinus rhythm
* Effective oral anticoagulation verified by International Normalized Ratio/INR (target > 2)
* QTc Bazett < 500 ms and PR < 280 ms on 12-lead ECG
* Completed treatment period with amiodarone (28 days ± 2 days)

Exclusion criteria:

Screening:

* Contraindication to oral anticoagulation
* Acute condition known to cause AF
* Permanent AF
* Paroxysmal AF
* Bradycardia < 50 bpm on the 12-lead ECG
* Clinically overt congestive heart failure:

  * with New York Heart Association (NYHA) classes III and IV heart failure
  * with LVEF < 35%
  * or NYHA class II with a recent decompensation requiring hospitalization or referral to a specialized heart failure clinic
  * or unstable hemodynamic conditions
* Severe hepatic impairment
* Previous treatment with class I or class III anti-arrhythmic drugs (including sotalol) if taken less than one week
* Previous history of amiodarone intolerance or toxicity
* Any contraindication as per dronedarone and amiodarone labelling
* Wolff-Parkinson-White Syndrome
* Previous ablation for atrial fibrillation or any planned ablation in the next 2 months
* Contraindicated concomitant treatment:

  * Potent cytochrome P450 (CYP3A4) inhibitors
  * Use of drugs or herbal products that prolong the QT interval and known to increase the risk of Torsades de Pointes
  * Class I or III anti-arrhythmic drugs (including sotalol)

Randomization:

* Bradycardia < 50 bpm on the 12-lead ECG
* Clinically overt congestive heart failure:

  * with New York Heart Association (NYHA) classes III and IV heart failure
  * with LVEF < 35%
  * or NYHA class II with a recent decompensation requiring hospitalization or referral to a specialized heart failure clinic
  * or unstable hemodynamic conditions
* Severe hepatic impairment
* Previous treatment with class I or class III anti-arrhythmic drugs (including sotalol) if taken less than one week
* Patient in whom the following contraindicated concomitant treatment is mandatory:

  * Potent cytochrome P450 (CYP3A4) inhibitors
  * Use of drugs or herbal products that prolong the QT interval and known to increase the risk of Torsades de Pointes
  * Class I or III anti-arrhythmic drugs (including sotalol)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AF recurrences | one month after randomization
  two consecutives 12-lead ECG or Trans-Telephonic ECG monitoring (TTEM) approximatively 10 minutes apart and both showing AF

SECONDARY OUTCOMES:
AF recurrences | two months after randomization
Symptomatic bradycardia | two months after randomization
  Heart rate at rest < 50 beats per minute
Tachycardia | two months after randomization
  Heart rate at rest > 120 beats per minute
Dronedarone and amiodarone concentrations in plasma | 3 hours, 1 week, 2 weeks and 4 weeks after 1st Dronedarone intake
  Limited to a subset of countries

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (111):
- Australia (13):
  - Investigational Site Number 009, Adelaide
  - Investigational Site Number 013, Ballarat
  - Investigational Site Number 002, Garran
  - Investigational Site Number 007, Herston
  - Investigational Site Number 012, Hobart
  - Investigational Site Number 006, Liverpool
  - Investigational Site Number 010, Maroubra
  - Investigational Site Number 001, Nedlands
  - Investigational Site Number 004, New Lambton
  - Investigational Site Number 008, Redcliffe
  - Investigational Site Number 011, South Brisbane
  - Investigational Site Number 005, Southport
  - Investigational Site Number 003, Woolloongabba
- Austria (7):
  - Investigational Site Number 040-006, Braunau am Inn
  - Investigational Site Number 040-007, Innsbruck
  - Investigational Site Number 040-002, Linz
  - Investigational Site Number 040-001, Mödling
  - Investigational Site Number 040-005, Vienna
  - Investigational Site Number 040-003, Vienna
  - Investigational Site Number 040-004, Vienna
- Investigational Site Number 233001, Tallinn, Estonia
- Finland (4):
  - Investigational Site Number 246-001, Hyvinkää
  - Investigational Site Number 246-002, Hyvinkää
  - Investigational Site Number 246-004, Pori
  - Investigational Site Number 246-003, Seinäjoki
- France (10):
  - Investigational Site Number 250-006, Avignon
  - Investigational Site Number 250-009, Béziers
  - Investigational Site Number 250-002, Bron
  - Investigational Site Number 250-007, Cholet
  - Investigational Site Number 250-008, Lyon
  - Investigational Site Number 250-010, Nîmes
  - Investigational Site Number 250-003, Poitiers
  - Investigational Site Number 250-004, Toulouse
  - Investigational Site Number 250-005, Valence
  - Investigational Site Number 250-001, Vandœuvre-lès-Nancy
- Germany (11):
  - Investigational Site Number 276-003, Berlin
  - Investigational Site Number 276-006, Bernau
  - Investigational Site Number 276-001, Bonn
  - Investigational Site Number 276-011, Dresden
  - Investigational Site Number 276-010, Frankfurt am Main
  - Investigational Site Number 276-002, Hamburg
  - Investigational Site Number 276-008, Hamburg
  - Investigational Site Number 276-009, Heidenau
  - Investigational Site Number 276-004, Kiel
  - Investigational Site Number 276-005, Ludwigsburg
  - Investigational Site Number 276-007, Paderborn
- Israel (2):
  - Investigational Site Number 376002, Ashkelon
  - Investigational Site Number 376001, Beer Yaakov
- Italy (11):
  - Investigational Site Number 380-005, Ancona
  - Investigational Site Number 380-002, Barga
  - Investigational Site Number 380-004, Catania
  - Investigational Site Number 380-001, Como
  - Investigational Site Number 380-006, Cortona
  - Investigational Site Number 380-011, Mestre
  - Investigational Site Number 380-010, Palermo
  - Investigational Site Number 380-007, Roma
  - Investigational Site Number 380-003, Roma
  - Investigational Site Number 380-009, San Daniele del Friuli
  - Investigational Site Number 380-012, Varese
- Mexico (13):
  - Investigational Site Number 484017, Aguascalientes
  - Investigational Site Number 484012, Chihuahua City
  - Investigational Site Number 484008, Guadalajara
  - Investigational Site Number 484009, Guadalajara
  - Investigational Site Number 484015, Guadalajara
  - Investigational Site Number 484002, León
  - Investigational Site Number 484016, México
  - Investigational Site Number 484004, México
  - Investigational Site Number 484005, Monterrey
  - Investigational Site Number 484003, Monterrey
  - Investigational Site Number 484001, Querétaro
  - Investigational Site Number 484013, Saltillo
  - Investigational Site Number 484011, Tijuana
- Netherlands (5):
  - Investigational Site Number 528003, Amsterdam
  - Investigational Site Number 528005, Goes
  - Investigational Site Number 528002, Groningen
  - Investigational Site Number 528001, Maastricht
  - Investigational Site Number 528004, Rotterdam
- Portugal (2):
  - Investigational Site Number 620005, Amadora
  - Investigational Site Number 620001, Lisbon
- South Korea (6):
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410006, Suwon
- Spain (10):
  - Investigational Site Number 724008, A Coruña
  - Investigational Site Number 724004, El Palmar (murcia)
  - Investigational Site Number 724005, L'Hospitalet de Llobregat
  - Investigational Site Number 724003, Lleida
  - Investigational Site Number 724010, Madrid
  - Investigational Site Number 724001, Madrid
  - Investigational Site Number 724002, Majadahonda
  - Investigational Site Number 724006, Seville
  - Investigational Site Number 724007, Tarragona
  - Investigational Site Number 724009, Valencia
- Switzerland (2):
  - Investigational Site Number 756001, Basel
  - Investigational Site Number 756002, Sankt Gallen
- Taiwan (9):
  - Investigational Site Number 158006, Kaohsiung City
  - Investigational Site Number 158005, Kaohsiung Hsien,
  - Investigational Site Number 158004, Taichung
  - Investigational Site Number 158003, Taichung
  - Investigational Site Number 158009, Taichung
  - Investigational Site Number 158002, Taipei
  - Investigational Site Number 158001, Taipei
  - Investigational Site Number 158008, Taipei
  - Investigational Site Number 158007, Tao Yuan Hsien
- United Kingdom (5):
  - Investigational Site Number 826006, Belfast
  - Investigational Site Number 826-005, Bournemouth
  - Investigational Site Number 826-001, Carshalton
  - Investigational Site Number 826-002, Gloucester
  - Investigational Site Number 826-007, Wrexham

REFERENCES:
- [Derived] Naccarelli GV, Bhatt DL, Camm AJ, Le Heuzey JY, Lombardi F, Tamargo J, Martinez JM, Naditch-Brule L; ARTEMIS AF Investigators. Evaluation of the Switch From Amiodarone to Dronedarone in Patients With Atrial Fibrillation: Results of the ARTEMIS AF Studies. J Cardiovasc Pharmacol Ther. 2020 Sep;25(5):425-437. doi: 10.1177/1074248420926874. Epub 2020 Jun 5. PMID 32500725